CLINICAL TRIAL: NCT01717911
Title: ß-Cell Function and Glycemic Control of Basal Insulin, Metformin or Sitagliptin in Newly Diagnosed Type 2 Diabetic Patients With Moderate Hyperglycemia
Brief Title: ß-Cell Function and Glycemic Control in Newly Diagnosed Type 2 Diabetic Patients With Moderate Hyperglycemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Division of Endocrinology and Metabolism, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB 201007016MB; NSC-2314-B-075-014 (Other Grant/Funding Number: NSC-2314-B-075-014)
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes
Keywords: Newly diagnosed type 2 diabetes; Insulin, metformin, sitagliptin; beta-cell function, glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; Insulin, Isophane; Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Active Comparator): The titration of metformin was used 500 mg for an adjust unit in splitting dose with the same target to the maximum daily dose of 2550 mg (1000 mg twice daily and then 850 mg tid).
  Interventions: Drug: Metformin
- Sitagliptin (Experimental): The subjects treated with sitagliptin started with 100 mg before breakfast once daily. The dosage was fixed as 100mg per day. Decreased by 50mg if fasting blood glucose was <70mg /dl, discontinued the study if blood glucose was still <70mg/dl under sitagliptin 50mg per day.
  Interventions: Drug: Sitagliptin
- Insulin (Experimental): In the insulin therapy group (Insulin glargine), subjects were instructed in the techniques for insulin injection and home capillary glucose monitoring. Daily dose was administrated before breakfast.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — In the insulin therapy group (Humulin-N), subjects were instructed in the techniques for insulin injection and home capillary glucose monitoring. Two third daily dose was administrated before breakfast and one third at bedtime. Insulin doses were titrated every 3 days to achieve target fasting plasma glucose values between 90 and 130 mg/dl.
  Other Names: Humulin-N
  Arms: Insulin
Drug: Metformin — The titration of metformin was used 500 mg for an adjust unit in splitting dose with the same target to the maximum daily dose of 2550 mg (1000 mg twice daily and then 850 mg tid).
  Other Names: Glucophage
  Arms: Metformin
Drug: Sitagliptin — The subjects treated with sitagliptin started with 100 mg before breakfast once daily. The dosage was fixed as 100mg per day. Decreased by 50mg if fasting blood glucose was <70mg /dl, discontinued the study if blood glucose was still <70mg/dl under sitagliptin 50mg per day.
  Other Names: Januvia
  Arms: Sitagliptin

SUMMARY:
We have found that a 6-month course of insulin therapy after a short-term intensive insulin therapy could shorten the period of hyperglycemia to preserve ß-cell function and further improve long-term glycemic control in recently diagnosed type 2 diabetes with severe hyperglycemia (>300 mg/dl, with HBA1C level around 9-11%) in our previous study. We thus hypothesized that a 6-month course of basal insulin therapy could also help to preserve ß-cell function in newly diagnosed type 2 diabetes with moderate hyperglycemia (200-300 mg/dl). This prospective study is outpatient-based to evaluate whether 6-month basal insulin therapy versus oral anti-diabetic treatment (Metformin and sitagliptin) soon after the diagnosis of type 2 diabetes with moderate hyperglycemia (200-300 mg/dl) is associated with better ß-cell function reservation. We skip a short-term intensive admission course of insulin therapy as our previous study in newly diagnosed type 2 diabetes with severe hyperglycemia.

DETAILED DESCRIPTION:
ß-Cell dysfunction and decreased insulin sensitivity are the main pathophysiological defects responsible for the development of hyperglycemia. There is a progressive deterioration in ß-cell function and mass in type 2 diabetics. Optimal metabolic control, especially early intensive glycemic control, plays a role in the prevention of progressive ß-cell dysfunction and possibly destruction of the ß-cells with worsening of diabetes.

We have found that a 6-month course of insulin therapy after a short-term intensive insulin therapy could shorten the period of hyperglycemia to preserve ß-cell function and further improve long-term glycemic control in recently diagnosed type 2 diabetes with severe hyperglycemia (>300 mg/dl, with HBA1C level around 9-11%) in our previous study. We thus hypothesized that a 6-month course of basal insulin therapy could also help to preserve ß-cell function in newly diagnosed type 2 diabetes with moderate hyperglycemia (200-300 mg/dl). This prospective study is outpatient-based to evaluate whether 6-month basal insulin therapy versus oral anti-diabetic treatment (Metformin and sitagliptin) soon after the diagnosis of type 2 diabetes with moderate hyperglycemia (200-300 mg/dl) is associated with better ß-cell function reservation. We skip a short-term intensive admission course of insulin therapy as our previous study in newly diagnosed type 2 diabetes with severe hyperglycemia.

This study also can assess what readily available parameter would predict which patients will achieve long-term successful glycemic control after correction of glucose toxicity.

Our results will provide evidence that a 6-month course of basal insulin therapy could shorten the exposure to moderate hyperglycemia and further improve beta-cell function to achieve long-term glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Recently diagnosed type 2 diabetic patients.
2. Fasting plasma glucose between 200-300 mg/dl (A1C level between 7% and 10%).
3. Those who age between 30 and 80 years old and can inject insulin by themselves.

Exclusion Criteria:

1. Previous treated with anti-diabetic medication
2. Pregnant or nursing women.
3. Impaired liver function (ALT > 120 U/L)
4. Impaired renal function (Serum creatinine >1.5 mg/dL in male, >1.4 mg/dL in female )
5. Recently suffered from MI or CVA.
6. Patients are acute intercurrent illness.
7. 2-hour C-peptide level < 1.8 ng/mL.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the comparison of A1C change. | Dec. 2013
  The primary outcome was the comparison of A1C change.

SECONDARY OUTCOMES:
Beta-cell function and insulin sensitivity and the proportion of subjects who reached the treatment target (A1C <7.0% or <6.5% at 6 months). | Dec 2013
  The secondary efficacy analysis was the beta-cell function and insulin sensitivity calculated from OGTT and the proportion of subjects who reached the treatment target (A1C <7.0% or <6.5% at 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Harn-Shen Chen, MD, Phd, Principal Investigator — Division of Endocrinology and Metabolism
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Chen HS, Wu TE, Jap TS, Hsiao LC, Lee SH, Lin HD. Beneficial effects of insulin on glycemic control and beta-cell function in newly diagnosed type 2 diabetes with severe hyperglycemia after short-term intensive insulin therapy. Diabetes Care. 2008 Oct;31(10):1927-32. doi: 10.2337/dc08-0075. Epub 2008 Jun 12. PMID 18556343